CLINICAL TRIAL: NCT00130702
Title: A Phase II Study of Iressa (Gefitinib), in Patients With Relapsed or Refractory Acute Myelogenous Leukemia and in Older Patients With Newly Diagnosed Acute Myelogenous Leukemia
Brief Title: Study of Iressa in Patients With Relapsed or Refractory Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Daniel J. DeAngelo, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-086
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Myelogenous Leukemia, Acute
Keywords: AML; acute myelogenous leukemia; gefitinib; Iressa
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefitinib (Iressa) (Experimental): All patients will receive Gefitinib (Iressa) at a dose of 750 mg orally (three 250 mg tabs) each day.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib — gefitinib (Iressa) at a dose of 750 mg, once per day
  Other Names: Iressa

SUMMARY:
The purpose of this study is to determine how effective, and to what extent, Iressa is in the treatment of acute myelogenous leukemia.

DETAILED DESCRIPTION:
Patients will receive Iressa daily until either disease progression or intolerable toxicity develops. On Day 1 of treatment, a physical exam and bloodwork will be performed. Once weekly for the first 8 weeks, a physical exam and complete blood count with differential will be performed.

For the first year, a physical exam, bloodwork will be performed monthly. Bone marrow biopsies will be performed after the first month of therapy and then every 3 months for the first year. After the first year a physical exam, bloodwork will be performed every 3 months and bone marrow biopsies every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically documented acute myelogenous leukemia and either not be a candidate for myelosuppressive chemotherapy due to age or comorbid disease; or have relapsed acute myelogenous leukemia or be refractory to standard therapy and not likely to require cytoreductive therapy within 30 days.
* ECOG performance status 0, 1 or 2
* Age > 18 years
* Adequate kidney and hepatic function
* Greater than 4 weeks from any chemotherapy, radiotherapy, immunotherapy, or systemic steroid therapy with the exception of hydroxyurea.
* Greater than 2 months following bone marrow or peripheral blood stem cell transplantation or donor lymphocyte infusion.

Exclusion Criteria:

* Uncontrolled active infection
* Urgent need for cytoreductive chemotherapy, surgery, or radiotherapy
* Current chemotherapy or chemotherapy within the last 4 weeks.
* Pregnancy or nursing mothers
* Infection with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of Iressa in patients with acute myelogenous leukemia

SECONDARY OUTCOMES:
To determine the safety of Iressa in patients with acute myelogenous leukemia | 2 years
to determine the biologic activity of Iressa in patients with acute myelogenous leukemia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States